CLINICAL TRIAL: NCT02473575
Title: Does a Commercial Caffeine Supplement Improve 5 km Run Performance in a Field Setting?
Brief Title: Does a Caffeine Gum Improve 5 km Run Performance in a Competition/Field Setting?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Principal Investigator, Tony Lynn, Senior Lecturer in Nutrition, Sheffield Hallam University
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: SBSREC1314/39
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Running Performance
Keywords: Caffeine, running, performance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Caffeine gum (Experimental): caffeine (300 mg) in gum form x 1 ingestion
  Interventions: Dietary Supplement: caffeine gum
- Placebo gum (Placebo Comparator): placebo gum consumed x 1 ingestion
  Interventions: Dietary Supplement: placebo gum
- Non-intervention group (No Intervention): A third group of runners will be used to adjust for changes in environmental conditions. They will complete 2 runs without consuming either placebo or experimental treatment

INTERVENTIONS:
Dietary Supplement: caffeine gum — Gum is consumed 30 minutes before commencement of run
  Arms: Caffeine gum
Dietary Supplement: placebo gum — Gum is consumed 30 minutes before commencement of run
  Arms: Placebo gum

SUMMARY:
The purpose of this study is to determine whether caffeine gum improves the performance of runners completing free timed mass participation 5 km runs in the United Kingdom (UK)

DETAILED DESCRIPTION:
The study will investigate the ability of an acute intake of caffeine gum to improve performance in recreationally trained runners completing park runs. Park runs are free, timed 5 km mass participation running events that are held in a number of parks around the UK every Saturday morning.

A total of 60 recreationally trained runners will be recruited to the study. Of these, 30 will be assigned to a randomised placebo-controlled double-blind cross-over trial. The remaining 30 will be assigned to a non-intervention comparison group. The non-intervention group will be used to account for the effect of changing environmental conditions on running performance.

All participants will complete two 5 km park runs separated by no more than 2 weeks. Participants on the intervention study arms will consume either caffeine or placebo gum 30 minutes before they run. The order of consumption will be randomised. The caffeine gum will contain 300 mg (with an approximate 85% bioavailability). Participants will be asked to abstain from any caffeine containing beverages or food for 18 hours before each run. They will also be asked to record their dietary intake for the day before and the morning of the run and to repeat this for their second trial. Physical activity on the days leading up to each 5 km run will also be recorded and participants will be asked to closely replicate their activity in the week leading up to each trial. They will also be asked to keep training intensity and duration light during the 48 hours leading up to each trial.

The primary outcome measure will be change in overall time for the 5 km runs. Other outcome measures will be ratings of perceived exertion, 1 km split times and average heart rate.

The study size was calculated using an online software package (http://www.sportsci.org/resource/stats/), adopting a power of 80% and an alpha of 0.05. Using within-person standard deviation from runners completing a local parkrun and an expected effect size of 1.2% (Bridge and Jones (2006) J Sports Sciences. 24(4):433-9) a sample size of 25 runners was calculated for the intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult runners with evidence of having recently ran 5 km in under 25 minutes

Exclusion Criteria:

* Current musculoskeletal injury, history of adverse response to caffeine, presence or history of cardiovascular disease, heart rhythm disorders or hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in 5 km run time | calculated after 2nd run (runs separated by 7 days)
  The difference in finishing time on placebo v caffeine; recorded in seconds

SECONDARY OUTCOMES:
Change in ratings of perceived exertion (RPE) | calculated after 2nd run (runs separated by 7 days)
  The difference in RPE on placebo v caffeine; using a 6-20 Borg scale

OTHER OUTCOMES:
Change in pacing | calculated after 2nd run (runs separated by 7 days); placebo v caffeine
  1 km split times in sec will be recorded manually and overall pace using GPS (km/h)
Change in average heart rate | calculated after 2nd run
  Recorded in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lynn, PhD, Principal Investigator — Sheffield Hallam University
Locations (1):
- Sheffield Hallam University, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Lynn A, Shaw C, Sorsby AC, Ashworth P, Hanif F, Williams CE, Ranchordas MK. Caffeine gum improves 5 km running performance in recreational runners completing parkrun events. Eur J Nutr. 2024 Jun;63(4):1283-1291. doi: 10.1007/s00394-024-03349-3. Epub 2024 Feb 24. PMID 38400919